CLINICAL TRIAL: NCT03431662
Title: Computerized Tomography (CT) Scan Study of Bone Healing Following Open Wedge
Brief Title: Computerized Tomography (CT) Scan Study of Bone Healing Following Open Wedge Proximal Tibial Osteotomy
Acronym: CISKO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ellipse Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PR0251
Record Dates: First submitted 2017-07-20; First posted 2018-02-13 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Osteoarthritis; Varus Malalignment
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ellipse IM HTO Nail (Experimental): In this arm, the subjects varus malalignment is corrected with Ellipse Intramedullary High Tibial Osteotomy Intramedullary Nail, which is a CE device. The device achieves the correction via progressive distraction osteogenesis.
  Interventions: Procedure: Ellipse IM HTO Nail
- TomoFix (Active Comparator): In this arm, the subjects varus malalignment is corrected with Synthes TomoFix system, which is a CE device. The device achieves the correction via fixating an accute intraoperative correction of the varus malalignment.
  Interventions: Procedure: TomoFix

INTERVENTIONS:
Procedure: Ellipse IM HTO Nail — A CT scan will be performed at 3 and 6 months postoperatively to assess the healing of the osteotomy site. Endpoint is 6 months.
  Other Names: Computerized Tomography (CT) Scan
  Arms: Ellipse IM HTO Nail
Procedure: TomoFix — A CT scan will be performed at 3 and 6 months postoperatively to assess the healing of the osteotomy site. Endpoint is 6 months.
  Other Names: Computerized Tomography (CT) Scan
  Arms: TomoFix

SUMMARY:
The purpose of this study is to assess whether there is a difference between the TomoFix and Ellipse Intramedullary HTO Nail System in terms of bone regeneration in the tibial wedge by performing a CT-scan at 3 and 6-months postoperatively.

DETAILED DESCRIPTION:
Malalignment of the knee joint causes arthritis in later life. Currently there are three surgical ways to treat knee arthritis: total knee replacement, partial knee replacement, and high tibial osteotomy (HTO). The former two very much focus on treating the effect of malalignment, i.e. removing the arthritic joint. However, HTO addresses the cause of the arthritis, namely the joint malalignment. This preserves the patient's joint and it means that a patient will start using the unaffected part of the knee joint more.

HTO involves cutting a wedge out the tibia to correct the alignment of that bone with the knee joint, to redistribute load from the affected medial part to lateral part. To keep the tibia in the new position, a medical nail device is attached to keep it in place and allow new bone to regenerate within the wedge. Currently, the market leader for HTO is the TomoFix (by DePuySynthes company) plate and nail device. As the name suggests, TomoFix is fixed at surgery and therefore the change in bone angle cannot be changed afterwards. It does mean that patients can be weight-bearing on the affected leg soon after the HTO procedure. A new CE-marked device is being tested in an interventional trial; it is produced by Ellipse Technologies. This device is an extendable nail and inserted intramedullary; following surgery the nail is tend slowly extended over a period of time until the bone correction is satisfactory.

The CISKO imaging study will assess whether there is a difference between the TomoFix and Ellipse system in terms of bone regeneration in the tibial wedge by performing a CT-scan at 3 and 6 months post-operatively. This will be quantified by two independent radiological reports. A secondary objective is to investigate patient satisfaction and also patient pain levels at these time intervals. The degree of bone healing is usually the main factor holding clinicians back when it comes to advising patients on what activities they can return to post-operatively. A difference in bone healing between the two systems may impact on the advice clinicians can give patients regarding recommencing more intense activities such as recreational sports, which ultimately could positively impact patients' health and well-being.

ELIGIBILITY:
Inclusion Criteria:

1. Indicated treatment with medial open wedge proximal tibial osteotomy, either with Tomofix device or Ellipse device
2. Provision of written informed consent
3. Males
4. Mental capacity

Exclusion Criteria:

1. Under age (< 18 years)
2. Patients lacking mental capacity.
3. Females
4. Current use of nicotine products.
5. Patients who cannot understand English and therefore cannot be consented.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Healing of the osteotomy site | 6-month postoperative
  Healing of the osteotomy site after final correction as assessed by two independent radiology reports based on visual assessment of the CT imaging. The scoring system is derived from a study by Brosset and colleagues (Brosset et al, 2011). In addition to a pure clinician perspective of the healing process, CT imaging data will also be used to quantify and describe:
  * definition of osteotomy line,
  * osteotomy margin,
  * osteotomy gap,
  * callus appearances,
  * callus to cortex ratio,
  * bridging of the bone, including complete union and healing.
  * application of region of interest (ROI) to quantify bone density of the callus formation

SECONDARY OUTCOMES:
Visual Analog Pain Scale | 6-month postoperative
  A patient reported outcome of their perception of pain
Osteotomy patient satisfaction questionnaire | 6-month postoperative
  A patient reported outcome of the patient's perception of satisfaction with treatment
SF-12 Quality of Life Questionnaire | 6-month postoperative
  A validated patient reported outcome.
KOOS Knee Health Questionnaire | 6-month postoperative
  A validated patient reported outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- North Cumbria University Hospitals NHS Trust, Carlisle, United Kingdom

IPD SHARING:
Plan to Share IPD: No